CLINICAL TRIAL: NCT06772636
Title: Effect of Music in Reducing Pain and Anxiety During Hysterosalpingography in Women With Primary Infertility: a Randomized Controlled Trial
Brief Title: Effect of Music in Reducing Pain and Anxiety During Hysterosalpingography in Women With Primary Infertility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MUSIC HSG
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music group (Experimental)
  Interventions: Procedure: music group
- non-music group (Other)
  Interventions: Procedure: non music group

INTERVENTIONS:
Procedure: music group — In the music group, the music chosen by the participant will be played through a speaker by the nursing staff during outpatient hysteroscopy. Music will be played through a speaker instead of headphones in order to maintain good communication and interaction between the participant and the doctor.
  Arms: music group
Procedure: non music group — Participants in the non-music group will undergo hysterosalpingography in the same setting and standard procedure without listening to any music.
  Arms: non-music group

SUMMARY:
This study aims to demonstrate the value of music in lowering pain and anxiety during hysterosalpingography in women with primary infertility

DETAILED DESCRIPTION:
This study aims to demonstrate the value of music in lowering pain and anxiety during hysterosalpingography in women with primary infertility

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years. Diagnosed with primary infertility (no prior pregnancy after at least 12 months of unprotected intercourse) and scheduled for HSG as part of infertility evaluation.

Exclusion Criteria:

* Using analgesics before or after the procedure, using antidepressants or sedative medications, being allergic to radio-opaque material, Current pregnancy or suspicion of pregnancy.Active pelvic inflammatory disease or history of severe pelvic infections within the last 6 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | 10 minutes
  Pain intensity will be assessed by visual analog scale during the procedure. visual analog scale ranging from 0 to 10 where 0 denotes no pain and 10 denotes maximum pain felt

SECONDARY OUTCOMES:
anxiety during procedure | 10 minutes
  anxiety will be measured using 10 cm VAS like score where 0 denotes no anxiety and 10 represents maximum anxiety

IPD SHARING:
Plan to Share IPD: Undecided